CLINICAL TRIAL: NCT00489008
Title: Phase II Stereotactic Body Radiotherapy for Stage I (T1-T2, N0, M0), Selective Stage II (Chest Wall T3, N0M0) or Isolated Peripheral Lung Recurrent Non-Small Cell Lung Cancer (NSCLC)
Brief Title: SRS Study in Patients With Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2005-0574; NCI-2012-01495 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2007-06-20; First posted 2007-06-21 (Estimated); Last update posted 2020-03-30 (Actual); Status verified 2020-03

CONDITIONS: Lung Cancer
Keywords: Lung Cancer; Non-Small Cell; Stereotactic Body Radiation Therapy; SBRT; NSCLC
MeSH Terms: conditions — Lung Neoplasms | interventions — Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Cohort 1 (Experimental): Stereotactic Body Radiation Therapy (SBRT) Stage I NSCLC
  Interventions: Procedure: Stereotactic Body Radiation Therapy (SBRT)
- Cohort 2 (Experimental): Stereotactic Body Radiation Therapy (SBRT) Selective Stage II NSCLC
  Interventions: Procedure: Stereotactic Body Radiation Therapy (SBRT)
- Cohort 3 (Experimental): Stereotactic Body Radiation Therapy (SBRT) Isolated Peripheral Lung Recurrent NSCLC
  Interventions: Procedure: Stereotactic Body Radiation Therapy (SBRT)

INTERVENTIONS:
Procedure: Stereotactic Body Radiation Therapy (SBRT) — Cohorts 1 & 2: 50 gray (GY) with 12.5 GY per Fraction for 4 treatments
  Cohort 3: 40 GY with 10 GY per Fraction for 4 treatments

SUMMARY:
The goal of this clinical research study is to learn if stereotactic body radiotherapy (SBRT) can help to control NSCLC. The safety of SBRT will also be studied.

Objectives:

To assess therapeutic efficacy and toxicities of stereotactic body radiotherapy (SBRT) for patients with medically inoperable stage I (T1-2, N0,M0), selective stage II (chest wall T3, N0M0) or isolated peripheral lung recurrent non-small cell lung cancer (NSCLC).

Primary goal: Improve 2 years progression free survival at the treated primary tumor site.

Secondary goals:

1. Improve disease free survival, disease specific survival and overall survival at 2 years.
2. Decrease grade 3 and above acute and/or chronic toxicities.
3. Collect blood for future biomarkers study

DETAILED DESCRIPTION:
Stereotactic body radiotherapy is designed to provide an image guided, more focused, dose escalated radiotherapy over a shorter time frame (1 week rather than 7 weeks) than conventional radiation therapy. The goal of SBRT is to improve tumor control while reducing the side effects.

If you are found to be eligible to take part in this study, you will receive daily SBRT for 4 days in a row over a 45 minute time period. During the treatment, you will lie still on a table for about 45 minutes per day in the same position. The machine will deliver the dose according to the plan developed by the doctor and the dose will be controlled by a computer.

During the treatment, you will be seen by a doctor and research nurse once a week to evaluate possible side effects. A physical exam and a medical history will be done at these visits.

You will be taken off study early if the disease gets worse or intolerable side effects occur.

You will have a follow-up visit 6 weeks after completion of radiotherapy to check for side effects. You will continue to have follow-up visits that will decrease in frequency over time. You will have imaging tests (chest CT or positron emission computed tomography (PET) scan) and routine blood tests (about 2 teaspoons) at these follow-up visits.

This is an investigational study. SBRT is FDA approved for the treatment of lung cancer. About 138 patients will take part in this study. All will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Cohort 1: Histologically or cytologically documented NSCLC.
2. Cohort 1: Inoperable stage IA (T1N0MO), IB (T2N0MO) and selective stage II (T3 due to chest wall involvement, N0M0). Patient refuses surgery is eligible. Secondary lung cancer is eligible if primary cancers have been cured or stable with life expectance longer than 2 years. If primary cancer is lung cancer, patient needs to be lung cancer free for more than 5 year for same histology or more than 2 years for different histology.
3. Cohort 1: Patients with hilar or mediastinal lymph nodes <= 1cm and no abnormal hilar or mediastinal uptake on PET will be considered N0. Patients with > 1 cm hilar or mediastinal lymph nodes on CT or abnormal PET (including suspicious but on-diagnostic uptake) may still be eligible if directed tissue biopsy of all abnormally identified areas are negative for cancer. Patient who received induction chemotherapy or other systemic therapy are eligible.
4. Cohort 1: Performance score Karnofsky performance status (KPS) 60-100.
5. Cohort 2: Histologically or cytologically documented NSCLC.
6. Cohort 2: Inoperable isolated lung parenchyma recurrent NSCLC without evidence of lymph node or mediastinal involvement (clinical stage T1-2, chest wall involvement T3, N0M0) after surgical resection or definitive radiotherapy with/without chemotherapy. Recurrent disease is defined as NSCLC with same histology, same lobe that recurs within 5 years after initial definitive therapy. Patient refuses surgery is also eligible. Patient received systemic therapy is eligible.
7. Cohort 2: Performance score KPS 60-100.
8. Cohort 3: Histologically or cytologically documented NSCLC.
9. Cohort 3: Previous history of NSCLC that has been cured or stable. New development of inoperable isolated lung parenchyma lesion that has been documented histologically or cytologically as NSCLC without evidence of lymph node or mediastinal involvement (clinical stage T1-2, chest wall involvement T3, N0M0) and not eligible for cohort 1 and recurrent disease as defined in Cohort 2. This includes NSCLC happens within 5 years after initial definitive treatment of prior NSCLC, and/or is located in the different lobes.
10. (cont.) Cohort 3: Possible stage IV disease is eligible as long as it meets the criteria above since there is no definitive way to confirm it. Patient refuses surgery is eligible. Patient received systemic therapy is eligible.
11. Cohort 3: Performance score KPS 60-100.

Exclusion Criteria:

1. Any tumor involving main bronchus, major vessels, heart, esophagus, trachea, carina, spinal cord.
2. Any tumor that causes collapsed lobe of lung.
3. Any tumor with malignant pleural effusion.
4. Direct evidence of hilar, mediastinal lymph node or distant metastasis based on staging work up.
5. Pregnancy. Patients (men and women) of child bearing potential should use an effective (for them) method of birth control throughout their participation in this study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 141 (Actual)
Dates: Start 2005-11-21 (Actual); Primary Completion 2017-06-02 (Actual); Study Completion 2017-06-02 (Actual)

PRIMARY OUTCOMES:
Progression Free Survival (PFS) at Treated Primary Tumor Site | 2 Years
  Progression free survival at the primary site evaluated by series CT of chest with contrast for every follow up (except 6 weeks after radiotherapy) for two years. PET information considered for calculation of PFS particularly for distant metastasis and/or additional lesions.
  Population proportion for two-year PFS estimated using Clopper-Pearson 95% confidence intervals.

CONTACTS AND LOCATIONS:
Overall Officials: Joe Y. Chang, MD, PhD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Sun B, Brooks ED, Komaki R, Liao Z, Jeter M, McAleer M, Balter PA, Welsh JD, O'Reilly M, Gomez D, Hahn SM, Sepesi B, Rice DC, Heymach JV, Chang JY. Long-Term Outcomes of Salvage Stereotactic Ablative Radiotherapy for Isolated Lung Recurrence of Non-Small Cell Lung Cancer: A Phase II Clinical Trial. J Thorac Oncol. 2017 Jun;12(6):983-992. doi: 10.1016/j.jtho.2017.02.018. Epub 2017 Mar 1. PMID 28259750
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org